CLINICAL TRIAL: NCT00272272
Title: The Nolwenn Effect in a Geriatric Nursing Home Setting
Brief Title: Fall Prevention in a Geriatric Nursing Home Setting Using the Music of Nolwenn Leroy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Primary Investigator, Carrick Institute for Graduate Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CI-01-01-06-01
Record Dates: First submitted 2006-01-03; First posted 2006-01-05 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Ataxia
Keywords: Fall Prevention, Music Therapy, Geriatric, Nursing Home
MeSH Terms: conditions — Ataxia | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balance and Music Listening (Experimental): Music therapy
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — Listening to Music while standing

SUMMARY:
Falls are the largest cause of death in the elderly and those with dementia have even a higher incidence of falling. The purpose of this study is to determine whether listening to the Music of Nolwenn Leroy is effective in fall prevention in those elderly patients who are residents in a Geriatric Nursing Home Facility. The music of Nolwenn Leroy has been shown to be effective in fall reduction in a different setting (Posturographic Changes and Fall Prevention associated with Music Therapy: The Nolwenn Effect (USA ClinicalTrials.gov Identifier: NCT00121693) )with results better than listening to Mozart of any other music.

DETAILED DESCRIPTION:
Falls are a serious health issue and are the greatest cause of death in the elderly. The use of the music of Nolwenn Leroy in fall prevention has been reported at a major scientific meeting Posturographic Changes and Fall Prevention associated with Music Therapy: The Nolwenn Effect (USA ClinicalTrials.gov Identifier: NCT00121693) featured at the 7th Annual American Music Therapy Association Conference in Orlando, Florida, Nov 15-20, 2005 and is in publication in the indexed literature. Decreasing falls in a geriatric nursing home setting is associated with the saving of lives. We propose the utilization of the Nolwenn Effect in our resident geriatric population and comparing fall rates to those we have carefully recorded in the past.

Daily listening to selections from Nolwenn Leroy's CD "Nolwenn" have been played for one month in the community gathering areas of our fourth floor dementia unit in the morning for approximately 5-10 minutes. This unit has an increased rate of falls due to the characteristics of its residents and our one month retrospective study has demonstrated a statistical reduction in the rate of falls subsequent to the daily listening of Nolwenn Leroy music. We propose to expand the listening of music to the entire building and study the Nolwenn Effect on the fall rate of all residents over the calendar year 2006.

Preliminary observations have been associated with a decrease rate of falls on our dementia floor when compared to our previous fall rates. Our nursing staff is well trained in fall reporting and will continue to do so in the manner previously established before implementation of this study. This study is dependant upon the utilization of fall statistics previously established at our institution. The incorporation of these statistics will allow us to demonstrate a cost effective method of reducing falls that might save lives, evoke societal change and act as a model for other Geriatric Nursing Home settings.

ELIGIBILITY:
Inclusion Criteria:

* Full time resident in Geriatric Facility

Exclusion Criteria:

* All others

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-12; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Changes in Fall rate | immediate pre and post balance testing

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD FACCN, Principal Investigator — Carrick Institute for Graduate Studies; Julie Kinney, MT-BC, Study Director — Carrick Institute for Graduate Studies; Elizabeth Eakes, MT-BC, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Budd Terrace Geriatric Nursing Home, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No